CLINICAL TRIAL: NCT05653102
Title: CR17-003 Truliant Knee PMCF: A Post-Market Domestic (US) and International Data Collection to Assess the Truliant Knee System
Brief Title: A Post-Market Domestic (US) and International Data Collection to Assess the Truliant Knee System
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR17-003
Record Dates: First submitted 2022-12-01; First posted 2022-12-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Prospective Subjects: Enrolled in the study pre-surgery. Subjects who agree to participate in the study that have not had surgery prior to being enrolled in the study.
  Interventions: Device: Truliant Total Knee System
- Retrospective to Prospective: Subjects enrolled in the study post- surgery then continue to participate in the study prospectively. Subjects who agree to participate in the study that have undergone surgery prior to enrollment in the study. Data for these subjects will collected from the subject's medical record for the time period prior to enrollment in the study containing data pertaining to the index surgery (retrospective data) and from the patient after they are enrolled in the study during the post-operative time period (prospectively).
  Interventions: Device: Truliant Total Knee System
- Retrospective Only Subjects: Subjects enrolled in the study post-study surgery with no intent to continue as prospective subjects. Patient's clinical record includes a signed HIPAA waiver allowing for the use of clinical record data for the purpose of clinical research outside of the operating institution.
  Interventions: Device: Truliant Total Knee System

INTERVENTIONS:
Device: Truliant Total Knee System — Total Knee Arthroplasty using Exactech's Truliant® branded components are compatible with Optetrak branded components.

SUMMARY:
A Post-Market Domestic (US) and International Data Collection to Assess the Truliant® Knee System

DETAILED DESCRIPTION:
Patient outcomes data is important for assessing the post-market safety and effectiveness of orthopedic medical devices. The purpose of this study is to collect clinical and patient outcomes and survivorship data for patients who have received or will receive a Truliant® knee prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA).

ELIGIBILITY:
Inclusion Criteria:

Cohort 1. Prospective / Subjects- Enrolled in the study pre-surgery

1. Subjects who agree to participate in the study that have not had surgery prior to being enrolled in the study.
2. Skeletally mature (18 years of age or older).
3. Subject is willing and able to provide written informed consent for participation in the study.
4. Subject is to receive a Truliant® total knee replacement for Osteoarthritis, Avascular Necrosis, Rheumatoid Arthritis, Post-Traumatic Arthritis, Polyarthritis, Primary Implantation Failure, or as a Conversion of Uni-Compartmental Knee.
5. The knee replacement will be performed by the investigator or a surgeon sub-investigator.
6. The devices will be used according to the approved indications.

Cohort 2. Retrospective to Prospective / Subjects enrolled in the study post- surgery then continue to participate in the study prospectively.

1. Subjects who agree to participate in the study that have undergone surgery prior to enrollment in the study. Data for these subjects will collected from the subject's medical record for the time period prior to enrollment in the study containing data pertaining to the index surgery (retrospective data) and from the patient after they are enrolled in the study during the post-operative time period (prospectively).
2. Skeletally mature (18 years of age or older).
3. Subject is willing and able to provide written informed consent for participation in the study.
4. Subject received a Truliant® total knee replacement for Osteoarthritis, Avascular Necrosis, Rheumatoid Arthritis, Post-Traumatic Arthritis, Polyarthritis, Primary Implantation Failure, or as a Conversion of Uni-Compartmental Knee.
5. The knee replacement was performed by the investigator or a surgeon sub-investigator.
6. The devices are/were used according to the approved indications.

   * Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria, and have a minimum of the following pre-operative, operative, and applicable postoperative data available in the subject's medical records, related to the Truliant® knee prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for data submission: Pre-Operative:

     o Demographic Data
     1. Gender
     2. Age at surgery
     3. Height/Weight
     4. Indication for surgery
     5. Prior Injuries/Surgeries on index knee
     6. Comorbidities
   * Operative:

     * Date of Surgery
     * Type of Surgery (Primary / Revision)
     * All component product information, including catalogue reference numbers
     * Adverse Event Information, if applicable

Cohort 3. Retrospective Only Subjects enrolled in the study post-study surgery with no intent to continue as prospective subjects. Note: No prospective data may be collected from a subject if they are enrolled under this cohort unless the subject is willing and able to provide written informed consent for participation in the study.

1. Skeletally mature at the time of the surgery (18 years of age or older).
2. The patient's clinical record includes a signed HIPAA waiver allowing for the use of clinical record data for the purpose of clinical research outside of the operating institution.
3. The patients clinical record includes a documented procedure that includes, or is related to, TKA with a Truliant® Knee system device.
4. The knee replacement was performed by the investigator or a surgeon sub-investigator.
5. The devices are/were used according to the approved indications.
6. Special consideration should be taken to ensure that these subjects meet all inclusion criteria, none of the exclusion criteria and have a minimum of the following pre-operative, operative, and applicable postoperative data available in the subject's medical records, related to the Truliant® knee prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA). Prior to inclusion in the study, the following details must be available for submission:

   * Pre-Operative:

     * Demographic Data
     * Gender
     * Age at surgery
     * Height/Weight
     * Indication for surgery
     * Prior Injuries/Surgeries on index knee
     * Comorbidities
   * Operative:

     * Date of Surgery
     * Type of Surgery (Primary / Revision)
     * All component product information, including catalogue reference numbers Adverse Event Information, if applicable

Exclusion Criteria:

* Patient was <18 years of age at time of surgery
* Patient does not meet indicated population for use criteria for this device
* Patient is pregnant
* Patient is a prisoner
* Patient has a physical or mental condition that would invalidate the results
* Patient is contraindicated for the surgery (e.g., metal allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Truliant® Femoral Components, Tibial Inserts, Patellar Component and Tibial Trays are indicated for use in skeletally mature individuals undergoing primary surgery for total knee replacement due to osteoarthritis, osteonecrosis, rheumatoid arthritis and/or post-traumatic degenerative problems. They are also indicated for revision of failed previous reconstructions where sufficient bone stock and soft tissue integrity are present.
  The Truliant® Cemented Femoral Components, Tibial Inserts, Patellar Component and Tibial Trays are indicated for cemented use only. The Truliant® Porous Femoral Components are indicated for cemented or cementless use. The Truliant® Porous Tibial Trays are indicated for cemented or cementless use.
  Patients must qualify for surgery per indications and contraindications as well as meet all of the inclusion criteria and none of the exclusion criteria. The decision to offer a patient enrollment in this study is left to the discretion of the surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2035-01-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | Preoperative
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 1 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 2 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 3 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 4 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 5 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 6 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 7 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 8 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 9 year
  KOOS JR. - validated outcome score
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement JR. | 10 year
  KOOS JR. - validated outcome score
Oxford Knee Score | Preoperative
  OKS - validated outcome score
Oxford Knee Score | 1 year
  OKS - validated outcome score
Oxford Knee Score | 2 year
  OKS - validated outcome score
Oxford Knee Score | 3 year
  OKS - validated outcome score
Oxford Knee Score | 4 year
  OKS - validated outcome score
Oxford Knee Score | 5 year
  OKS - validated outcome score
Oxford Knee Score | 6 year
  OKS - validated outcome score
Oxford Knee Score | 7 year
  OKS - validated outcome score
Oxford Knee Score | 8 year
  OKS - validated outcome score
Oxford Knee Score | 9 year
  OKS - validated outcome score
Oxford Knee Score | 10 year
  OKS - validated outcome score
Visual Analog Scale (VAS) - Pain | Preoperative
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 6-weeks
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 6-months
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 1 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 2 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 3 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 4 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 5 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 6 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 7 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 8 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 9 year
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Pain | 10 year
  Visual scale from 1-10 (high score is better)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado Health, Aurora, Colorado
  - Florida Research Associates, DeLand, Florida
  - Nevada Orthopaedic and Spine Center, Las Vegas, Nevada
  - Crystal Clinic, Akron, Ohio
  - Medical University South Carolina, Charleston, South Carolina

REFERENCES:
- [Result] Meftah M, White PB, Ranawat AS, Ranawat CS. Long-term results of total knee arthroplasty in young and active patients with posterior stabilized design. Knee. 2016 Mar;23(2):318-21. doi: 10.1016/j.knee.2015.10.008. Epub 2016 Jan 29. PMID 26833096
- [Result] Scott CE, Clement ND, MacDonald DJ, Hamilton DF, Gaston P, Howie CR, Burnett R. Five-year survivorship and patient-reported outcome of the Triathlon single-radius total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1676-83. doi: 10.1007/s00167-014-2922-8. Epub 2014 Mar 13. PMID 24623184
- [Result] Martin A, Quah C, Syme G, Lammin K, Segaren N, Pickering S. Long term survivorship following Scorpio Total Knee Replacement. Knee. 2015 Jun;22(3):192-6. doi: 10.1016/j.knee.2015.01.007. Epub 2015 Mar 26. PMID 25818502